CLINICAL TRIAL: NCT01527188
Title: A Randomized, Double-blind, Placebo-controlled, Dose Ranging Phase II Study to Assess the Efficacy and Safety of 100IR, 300IR and 500IR Sublingual Tablets of House Dust Mite Allergen for the Treatment of Allergic Rhinitis in an Environmental Exposure Chamber Model
Brief Title: Efficacy and Safety of 100IR, 300IR, 500IR Sublingual House Dust Mite Tablets in Allergic Rhinitis Environment Exposure Chamber Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO67.10
Record Dates: First submitted 2012-02-01; First posted 2012-02-06 (Estimated); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Allergic Rhinitis Due to House Dust Mite
Keywords: HDM; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 100 IR (Experimental): 100 IR house dust mites allergen extract tablet
  Interventions: Drug: 100 IR house dust mites allergen extract tablet
- 300 IR (Experimental): 300 IR house dust mites allergen extract tablet
  Interventions: Drug: 300 IR house dust mites allergen extract tablet
- 500 IR (Experimental): 500 IR house dust mites allergen extract tablet
  Interventions: Drug: 500 IR house dust mites allergen extract tablet
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 100 IR house dust mites allergen extract tablet — One sublingual tablet daily during 6 months
  Other Names: Sublingual immunotherapy tablet
  Arms: 100 IR
Drug: 300 IR house dust mites allergen extract tablet — One sublingual tablet daily during 6 months
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR
Drug: 500 IR house dust mites allergen extract tablet — One sublingual tablet daily during 6 months
  Other Names: Sublingual immunotherapy tablet
  Arms: 500 IR
Drug: Placebo tablet — One sublingual tablet daily during 6 months
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of 3 doses of sublingual house dust mite (HDM) tablets versus placebo in the change from baseline of rhinitis total symptom score during the allergen chamber challenge before and after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* history of HDM rhinitis allergy for > 1 year
* sensitized to D. pteronyssinus and/or D. farinae
* RTSS >= 6 at least 2 time points during allergen challenge session

Exclusion Criteria:

* co sensitization to other allergen than HDM
* FEV1 < 80%
* Asthma GINA > 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 355 (Actual)
Dates: Start 2010-12-08 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, FRCPC, Principal Investigator — Cetero Research / PRACS Institute
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada

REFERENCES:
- [Derived] Worm M, Demoly P, Okamoto Y, Vidal C, Daghildjian K, Yan K, Casale TB, Bergmann KC. Safety of 300IR house dust mite sublingual tablet from pooled clinical trial and post-marketing data. World Allergy Organ J. 2024 Jun 25;17(7):100924. doi: 10.1016/j.waojou.2024.100924. eCollection 2024 Jul. PMID 39035788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 08 DEC 2010, Last Patient Last Visit 19 SEP 2012
Period: Overall Study
Arm/Group | 100 IR | 300 IR | 500 IR | Placebo
Started | 89 | 86 | 93 | 87
Completed | 75 | 68 | 70 | 75
Not Completed | 14 | 18 | 23 | 12
Not completed — Adverse Event | 5 | 5 | 11 | 0
Not completed — Withdrawal by Subject | 3 | 6 | 4 | 4
Not completed — Any other reason not above-mentioned | 6 | 7 | 8 | 8

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all randomized patients who received at least one dose of Investigational Product.
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 IR | 300 IR | 500 IR | Placebo | Total
Number analyzed (Participants) | 89 | 86 | 93 | 87 | 355
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.43 (10.089) | 32.53 (8.558) | 32.76 (9.327) | 31.25 (8.753) | 32.25 (9.190)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 45 | 44 | 47 | 183
  Male | 42 | 41 | 49 | 40 | 172

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End-of-treatment Period in the Area Under the Curve of the Rhinitis Total Symptom Score Recorded During 4 Hours (0-4h) of the Allergen Challenge
Description: The primary efficacy endpoint was the change from baseline (ChBL) (that is the first allergen challenge before treatment initiation) to the end-of-treatment period (6 months) in the Area Under the Curve (AUC) of the Rhinitis Total Symptom Score (RTSS) recorded during the four hours of the allergen challenge in the Environmental Exposure Chamber (EEC).
  The RTSS is the sum of four individual nasal symptom scores (rhinorrhoea, nasal congestion, nasal pruritus and sneezing), each assessed on a 0-3 rating scale. The RTSS was evaluated every 15 minutes in the first 2 hours and every 30 minutes in the last two hours, i.e. at 13 timepoints during each allergen challenge (from T0 to T240), and the scores were plotted against time (0 to 4 hours) to calculate the area under the curve, AUCRTSS_0-4h. A decrease in the AUCRTSS_0-4h value represents relief from the HDM allergic symptoms.
Time Frame: 6 months
Population: Full Analysis Set (FAS): all patients who received at least one dose of the investigational product.
  (Number of patients at Visit 7 for whom data is available).
Measure: Least Squares Mean (Standard Error); unit: RTSS * hour
Arm/Group | 100 IR | 300 IR | 500 IR | Placebo
Number analyzed (Participants) | 75 | 68 | 70 | 75
RTSS * hour | -715.83 (67.261) | -769.21 (70.659) | -795.58 (69.877) | -597.40 (67.401)
Statistical Analysis 1: Comparison: 500 IR vs Placebo; Test type: Superiority or Other; p = 0.0427, ANCOVA; Difference in LS Means = -198.18, 95% CI 2-sided [-389.82 to -6.55]
Statistical Analysis 2: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.0793, ANCOVA; Difference in LS Means = -171.82, 95% CI [-363.87 to 20.24]
Statistical Analysis 3: Comparison: 100 IR vs Placebo; The statistical test is not applicable due to the step-down approach performed to address the multiplicity issue; Test type: Superiority or Other; ANCOVA; Difference in LS Means = -118.43, 95% CI 2-sided [-305.90 to 69.04]

2. Secondary Outcome: Change From Baseline to the End-of-treatment Period in the Area Under the Curve of the Rhinitis Total Symptom Score Recorded During 2 Hours (2-4h) of the Allergen Challenge
Description: Change from baseline (ChBL) (that is the first allergen challenge before treatment initiation) to the end-of-treatment period (6 months) in the Area Under the Curve (AUC) of the Rhinitis Total Symptom Score (RTSS) recorded during the last two hours (2-4h) of the allergen challenge in the Environmental Exposure Chamber (EEC).
  The RTSS is the sum of four individual nasal symptom scores (rhinorrhoea, nasal congestion, nasal pruritus and sneezing), each assessed on a 0-3 rating scale.
Time Frame: 6 months
Population: Full Analysis Set (FAS): all patients who received at least one dose of the investigational product
Measure: Least Squares Mean (Standard Error); unit: RTSS * hour
Arm/Group | 100 IR | 300 IR | 500 IR | Placebo
Number analyzed (Participants) | 75 | 68 | 70 | 75
RTSS * hour | -390.34 (40.355) | -421.39 (42.400) | -424.77 (41.890) | -299.16 (40.430)
Statistical Analysis 1: Comparison: 500 IR vs Placebo; Test type: Superiority or Other; p = 0.0323, ANCOVA; Difference in LS Means = -125.61, 95% CI [-240.53 to -10.69]
Statistical Analysis 2: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.0376, ANCOVA; Difference in LS Means = -122.23, 95% CI [-237.38 to -7.08]
Statistical Analysis 3: Comparison: 100 IR vs Placebo; Test type: Superiority or Other; p = 0.1119, ANCOVA; Difference in LS Means = -91.18, 95% CI [-203.74 to 21.38]

ADVERSE EVENTS:
Time Frame: 6 months.
Description: Treatment-emergent adverse events (TEAEs) were defined as any AEs that started on or after the first administration of the investigational product and up to 30 days after the last administration of the investigational product.
Arm/Group | 100 IR | 300 IR | 500 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 1/89 | 1/86 | 2/93 | 0/87
Other Adverse Events (participants affected / at risk) | 82/89 | 73/86 | 81/93 | 71/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 IR (N=89) | 300 IR (N=86) | 500 IR (N=93) | Placebo (N=87)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 IR (N=89) | 300 IR (N=86) | 500 IR (N=93) | Placebo (N=87)
Oral pruritus (Gastrointestinal disorders) | 23 | 30 | 29 | 7
Oedema mouth (Gastrointestinal disorders) | 16 | 19 | 20 | 0
Nausea (Gastrointestinal disorders) | 12 | 8 | 7 | 4
Paraesthesia oral (Gastrointestinal disorders) | 3 | 3 | 6 | 1
Lip oedema (Gastrointestinal disorders) | 1 | 3 | 9 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 5 | 1 | 1 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 28 | 32 | 37 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 8 | 5
Ear pruritus (Ear and labyrinth disorders) | 19 | 21 | 23 | 8
Eye pruritus (Eye disorders) | 7 | 4 | 6 | 6
Headache (Nervous system disorders) | 29 | 22 | 29 | 38
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 4 | 4 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3 | 3 | 2
Lip pruritus (Gastrointestinal disorders) | 3 | 4 | 5 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 5 | 1 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 3 | 5 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 28 | 28 | 26 | 34
Pharyngitis (Infections and infestations) | 3 | 2 | 9 | 2
Chest discomfort (General disorders) | 7 | 4 | 3 | 3
Fatigue (General disorders) | 4 | 5 | 1 | 3
Pyrexia (General disorders) | 5 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 4 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 6
Forced expiratory volume decreased (Investigations) | 7 | 7 | 4 | 4
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 30 | 18 | 20 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 11 | 7 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 13 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 5 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No